CLINICAL TRIAL: NCT00539578
Title: A Double-Blind, Mulitcenter, Placebo-Controlled, Flexible-Dose Replicate Study of MK0777 Gel Extrusion Module (GEM) 3 mg B.I.D. to 8 mg B.I.D. in the Treatment of Outpatients With Generalized Anxiety Disorder
Brief Title: Treatment of Patients With Anxiety Disorder (0777-022)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0777-022; MK0777-022; 2007_622
Record Dates: First submitted 2007-10-01; First posted 2007-10-04 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0777 — Duration of Treatment: 4 weeks
Drug: Comparator: placebo (unspecified) — Duration of Treatment: 4 weeks

SUMMARY:
The purpose of the study is to examine the safety and efficacy of MK0777 during treatment for Generalized Anxiety Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ages 18 to 70

Exclusion Criteria:

* Women who are breastfeeding or pregnant
* Positive result at prestudy on urine drug screen for illicit drugs
* History of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2002-09; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC